CLINICAL TRIAL: NCT00327132
Title: Multicentre,Prospective Study of First-line Antibiotic Therapy for Early-stage Low-grade and High-grade Gastric Mucosa-associated Lymphoid Tissue-type Lymphoma and Potential Predicting Factor for Treatment Outcome
Brief Title: Prospective Study of First-line Antibiotic Therapy for Early-stage Gastric MALT Lymphoma for Treatment Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Tri-Service General Hospital (Other); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Changhua Christian Hospital (Other); Chi Mei Medical Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T3206
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Gastric MALT Lymphoma
Keywords: Early-stage Lg/Hg Gastric MALT Lymphoma; Eradication of Helicobacter pylori (Hp)
MeSH Terms: interventions — Omeprazole; Amoxicillin; Clarithromycin

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Drug: Omeprazole, Amoxicillin, Clarithromycin

INTERVENTIONS:
Drug: Omeprazole, Amoxicillin, Clarithromycin

SUMMARY:
1. The complete histological and molecular remission rate for antibiotics as 1st-line therapy for Hp-positive early-stage gastric lg- and hg-MALT lymphoma
2. The durability of complete histological remission after antibiotics
3. The usefulness of pattern of NF-kB and BCL-10 by IHC staining in prospectively predicting the Hp-dependence of gastric lg- and hg-MALT lymphoma
4. The frequency of t(11;18) translocation in gastric lg- and hg-MALT lymphoma in Taiwan.
5. The association between the CYP2C18/19 genetic polymorphisms and eradication of Hp infection after antibiotics.

DETAILED DESCRIPTION:
Background: Eradication of Helicobacter pylori (Hp) infection is well recognized as the initial therapy for early-stage low-grade gastric mucosa-associated lymphoid tissue-type lymphoma (lg-MALT lymphoma). On the other hand, high-grade transformed MALT lymphoma (hg-MALT lymphoma) is generally considered to arise from Hp-independent clones and thus to be unlikely to respond to antibiotic therapy. Our previous prospective studies have firstly demonstrated that 1st-line antibiotic therapy could achieve durable complete histological remission in two-third of Hp-positive stage IE hg-MALT lymphoma (Chen et al., J. Clin. Oncol., 2001), in which the long-term clinical outcomes were equivalent to those achievable in lg-MALT lymphoma (Chen et al. J Natl Cancer Inst, accepted). In addition, our laboratory studies have confirmed that t(11;18) translocation is associated with loss of Hp-dependence in lg-MALT lymphoma but infrequently found in high-grade tumors. We also found that nuclear translocation of NF-kB or BCL-10 (by immunohistochemical, IHC, staining) were useful markers to predict the Hp-dependence of both early-stage gastric hg- and lg-MALT lymphoma to antibiotic therapy (Kuo et al. JCO 2004 & Yeh et al. Blood 2005). In addition, recent data suggested cytochrome CYP2C18/19 genetic polymorphisms are associated with the metabolism of omeprazole, and thus the genotype of such enzymes might affect the efficacy of antibiotics for eradication of Hp infection.

Aims: A nationwide study to prospectively validate

1. The complete histological and molecular remission rate for antibiotics as 1st-line therapy for Hp-positive early-stage gastric lg- and hg-MALT lymphoma
2. The durability of complete histological remission after antibiotics
3. The usefulness of pattern of NF-kB and BCL-10 by IHC staining in prospectively predicting the Hp-dependence of gastric lg- and hg-MALT lymphoma
4. The frequency of t(11;18) translocation in gastric lg- and hg-MALT lymphoma in Taiwan.
5. The association between the CYP2C18/19 genetic polymorphisms and eradication of Hp infection after antibiotics.

Materials and Methods: Patients with newly, histologically proven stage IE / IIE-1 gastric lg- and hg-MALT lymphoma are eligible. Pre-treatment Hp infection status will be determined by histology, rapid urease test and serology. At time of registration, patients should agree to provide endoscopic biopsy specimen, including eight 4-mm histologic section for immunohistochemical study of NF-kB and BCL-10 and three 10-mm of section in eppendorf tube for RNA extraction and subsequent RT-PCR for t(11;18) translocation determination, which will be performed at the central laboratory. In addition, serum (from 5 mL of coagulated blood) as well as peripheral blood mononuclear cells (from 3 mL of heparized blood) will also collected before treatment for Hp-serology and CYP 2C18/19 genetic polymorphism detection, respectively. Hp-positive patients will receive 2-week of triple therapy, consisting of omeprazole, amoxicillin and clarithromycin (OAC regimen), and have first follow-up endoscopy 4 weeks later to determine the status of Hp infection and tumor response. Patients will then have sequential follow-up endoscopic examinations every 3 months until complete histological remission (CR) or disease progression; then every 6 months for complete responders. Patients with hg-MALT lymphoma who have stable or progressive disease after Hp eradication will immediately refer for systemic chemotherapy. CR was defined as regression of lymphoid infiltration to Wotherspoon's score <2 on all pathological sections of endoscopic biopsy specimens. The predictive value of NF-kB, BCL-10 and t(11;18) for complete histological remission after Hp eradication will be determined.

Expected Results: 1st-line antibiotic therapy will achieve complete histologic remission in 70-80% of Hp-positive stage IE gastric lg-MALT lymphoma and in 50-60% of stage IE hg-MALT lymphoma. The objective histologic CR rate in stage IIE-1 disease may be 30-40% for low-grade tumor and 20-30% for high-grade ones. The sensitivity and specificity of NF-kB and BCL-10 positive nuclear staining by IHC and of t(11;18) in predicting the Hp-independence will be both 80 - 90%. Ten - twenty per cent of enrolled patients will have CYP2C19 m1/m1, m1/m2 or m2/m2 genotypes (considered as omeprazole poor metabolizer), and they might have higher Hp eradication rate than those extensive metabolizers .

ELIGIBILITY:
Inclusion Criteria:

* The patients must have histologically confirmed primary gastric MALT lymphoma with or without clustering large cells (extranodal marginal zone lymphoma, and diffuse large cell lymphoma with features of MALT by REAL/WHO classification, Harris NL et al. 1994).

  * 1.1 The diagnosis of primary gastric lymphoma must fulfill the criteria of Dawson [38].

    * (1)No enlargement of peripheral or mediastinal lymph node;
    * (2)Peripheral blood smear revealing no leukemic or lymphomatous abnormalities;
    * (3)Predominant of alimentary tract lesions with any adenopathy corresponding to accepted lymphatic drainage route; and
    * (4)No involvement of liver or spleen except by extension of contiguous disease.
  * 1.2 The diagnosis of MALT lymphoma will be made by histopathologists from individual hospitals, in accordance with criteria defined by Isaacson et al. and Chang et al, and will be reviewed by the members of the TCOG Pathology Committee. This pathology review mechanism had been functioned well in the previous T1296 study (see J Natl Cancer Inst. 2005;97:1345-53)
  * 1.3 The patient must have no prior chemotherapy or radiotherapy for his/her gastric lg- or hg-MALToma.
* Patients must have evaluable disease by endoscopy and/or the nodal status by computed tomography. Endoscopic ultrasonography (EUS) is mandatory to evaluate the depth of tumor infiltration and for status of perigastric lymph node enlargement.
* Patients must have documented H. pylori infection before treatment, which will be evaluated by the following tests: histology, rapid urease test (CLO-test), C-13 urease breath test and serology.

  * 3.1 The following will be considered to have H. pylori infection: if any of above 4 tests show positive result.
* Patients must have either stage IE or IIE-1 disease, according to an adaptation of the Ann Abor staging system modified by Musshoff for primary extranodal lymphoma.

  * 4.1 Stage IE : lymphoma confined to the gastric wall without lymph node involvement.
  * 4.2 Stage IIE : localized involvement of one or more GI site(s) on one side of the diaphragm with lymph node involvement, any depth of lymphoma infiltration into the gut wall. 4.21 Stage IIE-1: involvement of perigastric lymph node. 4.22 Stage IIE-2: abdominal, but beyond perigastric, lymph nodal involvement.
* Patient must have signed the informed consent and agree to provide achieved pathologic material for immunohistochemical study and for RT-PCR t(11;18)(q21;q21) determination.

Exclusion Criteria:

* Patients with extensive gastrointestinal tract involvement are not eligible.
* Patients with previous history of extranodal lymphoma are not eligible.
* Patients with stage IIE-2 or beyond disease: infiltration of regional lymph node, e.g. paraaortic, renal hilar, retroperitoneal, mesenteric, or lymph node of gastrosplenic ligament and of hepatoduodenal ligament; or involvement of lymph node above and below diaphragm (Stage III) or other visceral organ involvement (stage IV) are not eligible.
* Patients with cardiopulmonary status that do not allow repeat endoscopy are not eligible.
* Patients with prior antibiotics, chemo- or radiotherapy for their gastric lymphoma are not eligible.
* Patients who had previous anti-H. pylori therapy and without pretreatment pathology achieve material for histological review and immunohistochemical study are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hp eradication rate and complete histological rate | 10 years

SECONDARY OUTCOMES:
overall survival (OS)Relapse-free survival (RFS) | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Town, Lin, M.D., PHD, Principal Investigator — Taiwan cooperative oncology group; Li Tzong Chen, M.D., Ph.D., Principal Investigator — Taiwan cooperative oncology group
Locations (5):
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Services General Hospital, Taipei

REFERENCES:
- See also: Related Info — http://english.nhri.org.tw/inst_cancer/ca_TCOG.php